CLINICAL TRIAL: NCT02230878
Title: A Randomized, Double-blind, Placebo-controlled Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of JNJ-42847922 in Healthy Male and Female Subjects
Brief Title: A Study to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-42847922 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR104154; 42847922EDI1003 (Other: Janssen-Cilag International NV); 2014-000600-95 (EudraCT Number)
Record Dates: First submitted 2014-08-14; First posted 2014-09-03 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
Keywords: JNJ-42847922; Phase 1; Healthy; Placebo
MeSH Terms: interventions — seltorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- JNJ-42847922, 5 milligram (mg) and Placebo (Experimental): Participants will be receive either 5 mg of JNJ-42847922 from Day 1 up to Day 10 or matching placebo from Day 1 up to Day 10.
  Interventions: Drug: JNJ-42847922 5 mg; Drug: Placebo
- JNJ-42847922, 10 mg and Placebo (Experimental): Participants will be receive either 10 mg of JNJ-42847922 from Day 1 up to Day 10 or matching placebo from Day 1 up to Day 10.
  Interventions: Drug: JNJ-42847922 10 mg; Drug: Placebo
- JNJ-42847922, 20 mg and Placebo (Experimental): Participants will be receive either 20 mg of JNJ-42847922 from Day 1 up to Day 10 or matching placebo from Day 1 up to Day 10.
  Interventions: Drug: JNJ-42847922 20 mg; Drug: Placebo
- JNJ-42847922, 40 mg and Placebo (Experimental): Participants will be receive either 40mg of JNJ-42847922 from Day 1 up to Day 10 or matching placebo from Day 1 up to Day 10.
  Interventions: Drug: JNJ-42847922 40 mg; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-42847922 5 mg — Participants will receive 5 mg of JNJ-42847922, from Day 1 up to Day 10.
  Arms: JNJ-42847922, 5 milligram (mg) and Placebo
Drug: JNJ-42847922 10 mg — Participants will receive 10 mg of JNJ-42847922, from Day 1 up to Day 10.
  Arms: JNJ-42847922, 10 mg and Placebo
Drug: JNJ-42847922 20 mg — Participants will receive 20 mg of JNJ-42847922, from Day 1 up to Day 10.
  Arms: JNJ-42847922, 20 mg and Placebo
Drug: JNJ-42847922 40 mg — Participants will receive 40 mg of JNJ-42847922, from Day 1 up to Day 10 .
  Arms: JNJ-42847922, 40 mg and Placebo
Drug: Placebo — Participants will receive matching placebo from Day 1 up to Day 10.

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, pharmacokinetic (the study of the way a drug enters and leaves the blood and tissues over time), dose-proportionality, accumulation, urinary excretion, pharmacodynamics (the study of how drugs act on the body) and sedative effects of JNJ-42847922 in healthy male and female participants.

DETAILED DESCRIPTION:
This is a Phase 1, double blind (a medical research study in which neither the researchers nor the participants know what treatment the participants is receiving), randomized (study drug assigned by chance), placebo controlled, multiple ascending dose study. The study will consist of 3 parts: a Screening period (Days -21 to -2), a Double-blind treatment period (Day -1 to Day 11), and a Follow-up period (within 7 to 14 days after last dose administration). In double blind treatment period, participants will be randomly assigned to 5, 10, 20, and 40 milligram (mg) or placebo. Number of participants with any clinically relevant changes (adverse events [AEs], laboratory results,electrocardiogram [ECG], Vital signs, Physical and neurological, sedation & concentration) and columbia suicide severity rating (CSSR) scale will be evaluated as primary outcome measure. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Women should not be of child bearing potential due to either tubal ligation or hysterectomy or who are postmenopausal (no spontaneous menses for at least 2 years
* Body Mass Index (BMI) between 18 and 30 kilogram per meter square (kg/m^2) inclusive (BMI=weight/height^2)
* Participants must be healthy / medically stable on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, retesting of an abnormal lab value(s) that may lead to exclusion will be allowed once during the screening phase
* Non-smokers (not smoked for 6 months prior to screening)
* Participant must be willing and able to adhere to the prohibitions and restrictions specified in this protocol

Exclusion Criteria:

* Clinically significant abnormal values for hematology, serum chemistry or urinalysis at screening or admission
* Clinically significant abnormal physical or neurological examination, vital signs or 12-lead electrocardiogram (ECG) at screening or admission
* History of or current significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematological disease, lipid abnormalities, bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, Parkinson's disease, infection, or any other illness that the Investigator considers should exclude the participant
* Serology positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies or human immunodeficiency virus (HIV) antibodies
* Subjects with a relevant history of a suicide attempt or suicidal behavior. Any recent suicidal ideation within the last 6 months (a level of 4 or 5), or who are at significant risk to commit suicide, as judged by the investigator using the columbia suicide severity rating score (C-SSRS)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Supine and Standing Systolic and Diastolic Blood Pressure (BP) | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
  BP is the pressure of the blood within the arteries. It is produced primarily by the contraction of the heart muscle. BP measurement is recorded by 2 numbers: systolic BP (SBP, BP when heart is contracting; it is the maximum arterial pressure during contraction of left ventricle) and diastolic BP (DBP, BP when heart is relaxing; it is the minimum arterial pressure during relaxation and dilation of ventricles).
Supine and Standing Heart Rate | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
Tympanic Temperature | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
12 Lead Electrocardiogram (ECG): RR, QRS, PR, QT, QTcB, QTcF Interval | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
Number of Participants with Adverse Events | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
Number of Participants With Change From Baseline in Laboratory Tests Results | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
  Laboratory values included Hematology, clinical chemistry and urinalysis.
Physical and Neurological Examination | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
  Physical and neurological examination will be performed.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (C[max]) | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
  The C(max) is the maximum plasma concentration which will be observed at the defined time points.
Time to Reach the Maximum Plasma Concentration (T[max]) | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
  The T[max] is time to reach the observed maximum plasma concentration.
Time to Reach Last Quantifiable Plasma Concentration (T[last]) | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
  The T[last] is time to reach the observed maximum plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to hour 24 Time (AUC [0-24]) | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
  AUC (0-24) is the area under the plasma concentration-time curve from time 0 to 24 hours post-dose.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-last]) | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
  AUC (last) is the area under the plasma concentration-time curve from time zero time of the last quantifiable concentration C(last), and C(last) is the last observed quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
  AUC (infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z), wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time; and C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Average Plasma Concentration at Steady-State (C[avg]) | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
  C(avg) is the average plasma concentration at steady state, calculated as AUC 0-24 divided by 24
Trough Plasma Concentration (C[trough]) | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
  Trough plasma concentration is the plasma concentration before dosing or at the end of the dosing interval of any dose other than the first dose.
Total Clearance (CL/F) | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
  CL/F is the total clearance of drug after extravascular administration, uncorrected for absolute bioavailability. It is calculated as Dose divided by AUC.
Volume of Distribution (Vd/F) | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
  Vd/F is the volume of distribution after extravascular administration, uncorrected for absolute bioavailability.
Elimination Half-life Period (t1/2) | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
  Elimination half-life associated with the terminal slope (lambda[z]) of the semi logarithmic drug concentration-time curve, calculated as 0.693/lambda (z).
Terminal slope (Lambda [z]) | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
  Terminal slope is defined by first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Mean Residence Time (MRT) | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
  MRT is the mean residence time calculated as area under the first moment curve at infinity (AUMC[0-∞]) divided by AUC[0-∞].
Amount of Drug Excreted in Urine (Ae) | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
  Ae is the amount of urine excreted in urine. It is calculated by multiplying the urinary volume with the urinary concentration.
Amount of Drug Excreted into Urine During the 24-hour Dosing Interval (Ae[0-24]) | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
  Ae(0-24h) is the amount of drug excreted into urine during the 24-hour dosing interval.
Percentage of Drug Excreted in Urine (Ae%dose) | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
  Ae%dose is the percentage of drug excreted into the urine calculated as (Ae divided by dose)∗100.
Renal Clearance (CL[R]) | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
  CL(R) is the renal clearance of the drug, calculated as Ae/AUC[0-infinity] on Day 1 or Ae(0-24)/AUC(0-24) on Day 5 and Day 10.

OTHER OUTCOMES:
Assessment of Sedation | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
  Sedation will be assessed using a reaction time (RT) test battery, the Critical Flicker Fusion (CFF) test and body sway.
Bond and Lader Visual Analogue Scale (B and L VAS) | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
  The B and L VAS includes 16 questions with VAS scales to rate subjective feelings.
Addiction Research Center Inventory Questionnaire (ARCI-49) | Baseline up to End of study (7-14 days after last dose) or Early withdrawal
  The ARCI-49 item questionnaire is developed specifically to measure subjective effects of drugs with diverse pharmacological actions.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (1):
- Berlin, Germany